CLINICAL TRIAL: NCT00979329
Title: Study on the Influence of Sunitinib and Sorafenib on Fatigue, Quality of Life and Depression in Patients With Metastatic Renal Cell Cancer or GIST
Brief Title: Study on the Influence of Sunitinib and Sorafenib on Fatigue, QoL, Depression in Patients With Metastatic RCC or GIST
Status: Completed | Type: Observational
Sponsor: Radboud University Medical Center (Other)
Responsible Party: Sponsor
Other Study IDs: UMCNONCO20082
Record Dates: First submitted 2009-09-17; First posted 2009-09-18 (Estimated); Last update posted 2017-11-28 (Actual); Status verified 2017-11

CONDITIONS: Renal Cell Cancer; Colorectal Cancer; GIST
Keywords: sunitinib; sorafenib; fatigue; depression; quality of life; metastatic RCC; colorectal cancer; GIST
MeSH Terms: conditions — Carcinoma, Renal Cell; Colorectal Neoplasms; Fatigue; Depression | interventions — Surveys and Questionnaires

STUDY DESIGN:
Observational Model: Case-Only | Time Perspective: Prospective
Oversight: Data Monitoring Committee: No

GROUPS / COHORTS (1):
- mRCC or GIST treated with sunitinib/sorafenib
  Interventions: Other: Questionnaires

INTERVENTIONS:
Other: Questionnaires — During the study three questionnaires must repeatedly be completed in by the patients: the BDI (PC) a depression scale, the EORTC-QLQ a quality of life assessment and the CIS20r, a fatigue scale and patients must fill in their medication on a list.

SUMMARY:
The purpose of this study is to assess the influence of Sunitinib and Sorafenib on fatigue, quality of life and depression in patients with metastatic renal cell or colorectal cancer or GIST. In order to get more insight in the mechanism of vascular endothelial growth factor (VEGF) related fatigue and if possible to come to a resolution for this side effect.

DETAILED DESCRIPTION:
When cure is not longer possible, cancer patients enter the palliative phase. For many types of cancer several treatment options are available. The goal of this treatment is to prolong survival, but maintenance or even improvement of quality of life is of equal importance. The currently available systemic treatment options consist of conventional cytotoxic therapy, hormonal therapy, immunotherapy and the so-called targeted therapies. Combinations of these therapies are also being used. Targeted therapy concerns the application of a new class of drugs that are specifically directed against one or more well-defined molecular targets that are relevant for carcinogenesis, cell cycle regulation, tumour progression, metastasis, tumour angiogenesis and/or apoptosis. Today, the most successful drugs in this class are directed against the vascular endothelial growth factor (VEGF) and the epidermal growth factor receptor (EGFR). There is an explosive development ongoing in this field and many new drugs become available that have new targets or inhibit a combinations of targets. Meanwhile, targeted therapy has shown efficacy in many types of cancer and is registered for several indications.

The toxicity profile of targeted therapies is still largely unknown, and the aetiology of many known side effects has not been clarified. This implies that the effective treatment of side effects is in an early phase of development. Given the impact of side effects on the quality of life of a patient, increased knowledge on this topic is urgently required. Currently only a few systematic studies are available that address this issue. At the moment, three targeted therapies that are directed against VEGF are registered and used in the Netherlands: Sunitinib (Sutent®) and Sorafenib (Nexavar ®) both oral drugs and Bevacizumab (Avastin®), an intravenously drug.

In this study we will focus on fatigue, quality of life and depression in patients with metastatic cancer, treated with Sunitinib and Sorafenib. Fatigue is one of the most frequent side effects of targeted therapy that are directed against VEGF and that can have a huge influence on the quality of life. The incidence of fatigue in patients using Sunitinib in phase I studies was 70% and the fatigue was often dose limiting. (1-4) In phase II-III studies the incidence was 27% - 51%. 5,6 In a phase III randomized, double-blind placebo-controlled trial of Sorafenib the incidence of fatigue in the Sorafenib group was 37% and in the placebo group 28%. (7) It is possible that fatigue is a symptom of depression or anxiety, alternatively, prolonged fatigue in itself can lead to depression or anxiety.8 There has been found a significant and positive correlation between anxiety and depressive symptoms and fatigue after treatment for cancer.

ELIGIBILITY:
Inclusion Criteria:

* patients with metastatic renal cell or GIST for whom treatment with Sunitinib or Sorafenib is planned
* Karnofsky score > 70%
* age > 18 year
* written informed consent for questionnaires

Exclusion Criteria:

* contra-indications for treatment with Sunitinib or Sorafenib
* patients who do not speak or write the Dutch language adequately
* previous systemic treatment within the last 7 days before start with the study, with Sunitinib, Sorafenib or Bevacizumab

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Study Population: patients with metastatic renal cell cancer or GIST who will be treated with Sunitinib or Sorafenib
Sampling Method: Non-Probability Sample
Enrollment: 100 (Actual)
Dates: Start 2008-05; Primary Completion 2011-12 (Actual); Study Completion 2015-12 (Actual)

CONTACTS AND LOCATIONS:
Overall Officials: C.M.L. van Herpen, MD, Phd, Principal Investigator — UMCN st Radboud
Locations (1):
- University Medical Center Nijmegen st Radboud, Nijmegen, Netherlands